CLINICAL TRIAL: NCT01329510
Title: The Effects of Methylphenidate on Sleep Patterns in Adults With ADHD: An Open Label Polysomnographic Study
Brief Title: Sleep and Nocturnal Melatonin in Adults With Attention Deficit Hyperactivity Disorder (ADHD)
Acronym: ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Dr. Shpirer Itzhak, Sleep & Snoring Clinic, Assaf Harofeh Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 106/05
Record Dates: First submitted 2010-09-01; First posted 2011-04-06 (Estimated); Last update posted 2011-04-06 (Estimated); Status verified 2005-08

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD; Adult
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- methylphenidate (Experimental)
  Interventions: Device: One-night polysomnographic recordings

INTERVENTIONS:
Device: One-night polysomnographic recordings — One-night polysomnographic recordings before and during methylphenidate treatment.

SUMMARY:
This study will investigate the effects of methylphenidate on sleep in adults with Attention Deficit/ Hyperactivity Disorder (ADHD) using polysomnographic parameters.

DETAILED DESCRIPTION:
Previous studies in children with Attention Deficit/ Hyperactivity Disorder (ADHD) have described the effect of stimulants on sleep patterns. However the data on adults with ADHD is sparse.

The aim of this study is to investigate the effects of methylphenidate on sleep in adults with ADHD using polysomnographic parameters.

ELIGIBILITY:
Inclusion Criteria:

* ADHD according to DSM-IV Criteria
* Positive ASRS questionnaire

Exclusion Criteria:

* Brain damage
* Brain encephalopathy
* Borderline IQ
* Affective disorder

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2005-08; Primary Completion 2006-12 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
polysomnographic parameters | one- night (day 1)

SECONDARY OUTCOMES:
sleep questionnaire | one week
  mini sleep questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Michael Khaigrekht, MD, Study Director — Memory, Attention And Learning Disabilities Unit, Assaf Harofeh Medical Center; Ran Shorer, M.A., Study Director — Memory, Attention And Learning Disabilities Unit, Assaf Harofeh Medical Center; Martin Rabey, MD, Study Director — Neurology Department , Assaf Harofeh Medical Center; Itzhak Shpirer, MD, Principal Investigator — Sleep And Snoring Clinic, Assaf Harofeh Medical Center; Shoky Shavit, M.A, Study Director — Memory, Attention And Learning Disabilities Clinic, Assaf Harofeh Medical Center
Locations (1):
- Assaf Harofeh Medical Center, Zrifin, Zrifin, Israel